CLINICAL TRIAL: NCT07371702
Title: PERsonalized Mammographic Screening in Norway; Additional Examination for Women With Increased Risk of Breast Cancer
Brief Title: PERsonalized Mammographic Screening in Norway
Acronym: PERMS
Status: Not yet recruiting | Type: Observational
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: Norwegian Cancer Society (Other); University Hospital, Akershus (Other); Oslo University Hospital (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 585149
Record Dates: First submitted 2026-01-05; First posted 2026-01-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Mammographic Breast Density; Risk Stratification
Keywords: Breast Cancer Screening; personalized screening; breast cancer screening; personalized screening
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women attending mammographic screening at three sites in BreastScreen Norway: Those 3-5% with the highest mammographic density in Study A and those with a false positive screening result in Study B will be offered additional imaging with digital breast tomosynthesis within 6 months after the screening examination (A) and an additional standard screening examination after one year (B)

SUMMARY:
The aim of this study is to assess attendance among women invited to additional breast imaging because they were identified as having an increased risk of breast cancer at screening. High-risk women were defined in two studies: Study A; women with high mammographic density, representing approximately 3-5% of screened women, and Study B; women with a false-positive screening result. Women in Study A will be offered an additional screening examination with digital breast tomosynthesis immediately within 6 months after the screening examination. Women in Study B will be offered an additional standard digital mammography examination one year after their initial screening.

ELIGIBILITY:
Inclusion Criteria:

* invited to screening
* extremely dense breast (Study A) or a false positive screening result (Study B)

Exclusion Criteria:

* Opted out or not signed written consent related to the study
* Women who have opted out from giving us permission to use screening data for quality assurance and research

Ages: 50 Years to 71 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women are invited to mammographic screening
Study Population: Study A will take place at the University Hospital of Akershus, while Study B will take place in Drammen, Vestre Viken Hospital and Oslo University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Attendance rate to extra imaging with digital breast tomosynthesis for women with extremely high mammographic density | Women will be invited to the extra examination with DBT within 6 months after index screening mammography.
  Women with extremely dense breasts will be offered an extra examination with DBT within 6 months after index screening mammography. The investigators will assess the attendance rate to this extra examination.
Attendance rate to an additional screening mammography for women with false positive screening result | Women will be invited to the additional screening mammography within 12 months after index screening mammography.
  Women with false positive screening result will be offered an additional screening mammography within 12 months after index screening mammography. The investigators will assess the attendance rate to this additional examination.

IPD SHARING:
Plan to Share IPD: No
Data will not be shared outside the project group